CLINICAL TRIAL: NCT03480113
Title: A Pilot Study of the Effectiveness of Mindfulness-based Intervention on Smoking Cessation: a Workplace Health-promoting Program
Brief Title: The Effectiveness of Mindfulness-based Intervention on Smoking Cessation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: Changhua Christian Hospital (Other)
Responsible Party: Principal Investigator, Yeh, professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS16175
Record Dates: First submitted 2018-03-14; First posted 2018-03-29 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-based Intervention (Experimental): 1 session of health education regrading the harms from smoking and 6 sessions of Mindfulness-based intervention, 1 hour each session.
  Interventions: Behavioral: Mindfulness-based Intervention
- Physical Fitness intervention (Active Comparator): 1 session of health education regrading the harms from smoking and 6 sessions of physical fitness and stretch exercise, 1 hour each session.
  Interventions: Behavioral: Physical fitness intervention

INTERVENTIONS:
Behavioral: Mindfulness-based Intervention — mindful breath, body scan, sitting meditation and walking meditation and so on.
  Arms: Mindfulness-based Intervention
Behavioral: Physical fitness intervention — giving the lessons of stretch exercise, aerobics to strength muscle and lung fuctions.
  Arms: Physical Fitness intervention

SUMMARY:
The present study will carry out a workplace health promotion via MBI to help smoking workers to quit smoking.

DETAILED DESCRIPTION:
The present study will carry out a workplace health promotion via MBI to help smoking workers to quit smoking. The study will adopt a longitudinal research design with randomized quasi-experimental trial. The smoking workers will recruited and be randomly assigned to Group A (one lesson of health education on smoking cessation and six lessons of MBI) or Group B (one lesson of health education on smoking cessation and six lessons of physical fitness). There will be 50 participants in each group. Data will be collected five times.

ELIGIBILITY:
Inclusion Criteria:

* volunteered employees with heavy smoker
* Full-time paid workers

Exclusion Criteria:

* Age < 20y or > 65y
* Part-time workers
* The workers are not willing to take part in the study

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Nicotine dependence level | Up to 8 months
  Fagerstrom Dependence Questionnaire was adopted to assess the level of Nicotine dependence

SECONDARY OUTCOMES:
Self-reported stress | Up to 8 months
  10 items of Perceived Stress Scale was adopted to assess the level of perceived stress. This scale uses the Likert five-point scoring method, from 0-4. The higher scores indicate higher pressure levels.
Psychological distress | Up to 8 months
  Psychological distress was measured by the Chinese Health Questionnaire (CHQ-12), a well-validated instrument. A total of 12 items using the Likert four-point scoring method, with scores ranged from 0-36. The higher scores indicates higher level of psychological distress.
the Level of mindfulness | Up to 8 months
  Measuring the level of Mindfulness, using the Likert five-point scoring method, a total of 39 questions, including the five concepts, namely: awareness (8 questions), description (8 questions), non-judging (8 questions), observation (8 questions), and non-reaction (7 questions). The higher scores indicate higher levels of mindfulness.
the level of CO | Up to 8 months
  The Smokerlyzer was adopted to assess the participants' CO level. <5ppm indicates nonsmoker; 5~7ppm indicates lighter smokers; ≧8ppm indicates heavy smokers.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Ling Huang, PhD, Principal Investigator — Department of Psychology, Chung Shan Medical University
Locations (1):
- AIDC, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No